CLINICAL TRIAL: NCT02690636
Title: Conventional Versus Hypofractionated Adjuvant Radiotherapy in Node Positive Breast Cancer. Phase III, Open Label, Randomized Trial. Comparing Local Control, Cosmetic Outcome, Arm Lymph Edema and Health Economic Perspectives
Brief Title: Conventional Versus Hypofractionated Radiotherapy in Node Positive Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Collaborators: Mit Ghamr Oncology Center (Other); Clinical Oncology department. Elmansoura University. (Unknown); Zagazig University (Other Government); Assiut University (Other); Tanta University (Other); Al-Azhar University (Other); Medical Research Institute. Department of Cancer Management and Research. (Unknown); Cairo University (Other); Clinical Oncology Department. Banha University. (Unknown); Ayadi El Mostakbal Cancer Center. Alexandria. (Unknown)
Responsible Party: Principal Investigator, Mahmoud Ellithy, Associate professor of clinical oncology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cure and More3
Record Dates: First submitted 2016-01-29; First posted 2016-02-24 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional (Active Comparator): The patients will receive adjuvant radiotherapy conventionally fractionated 5000 cgy fractionated by 200cgy daily fractions, five fractions per week over 5 weeks with an additional 200cgy daily for five days as boost for patients with breast conservative surgery.
  Interventions: Radiation: radiotherapy
- Hypofractionated (Experimental): The patients will receive adjuvant radiotherapy hypofractionated 266cgy daily fractions, five fractions per week for total 16 fractions and an additional five daily fractions will be added as boost for patients with breast conservative surgery.
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — daily fractions, five fractions per week.

SUMMARY:
Breast cancer patients operated with modified radical mastectomy or breast conservative surgery will be randomized for either adjuvant conventional radiotherapy versus hypofractionated radiotherapy for chest wall and axilla or breast and axilla.

The patients will be recruited for one year and will be followed for 5 years by monitoring local recurrence, cosmetic outcomes, health economic perspectives, and arm lymph edema.

DETAILED DESCRIPTION:
The investigators hypothesize that hypofractionated radiotherapy in node positive breast cancer is equally effective and safe as conventional fractionated radiotherapy. Breast cancer patients with pathological positive lymph nodes (N1 - N2) operated with modified radical mastectomy will be randomized 1:1 and also those with breast conservative surgery with positive lymph nodes will be randomized 1:1 for receiving either adjuvant conventional radiotherapy 200cgy x 25 fractions with 200cgy x 5 fractions boost for those with intact breast versus hypofractionated radiotherapy 266cgyx16 fractions and 266 cgy x 4 fractions boost for those with intact breast. The patients will be followed for 5 years to monitor locoregional recurrence, cosmetic outcomes, ipsilateral arm lymph edema. Health economic perspectives will be monitored by calculating cost effective analysis for both treatment plans.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG. (Eastern Cooperative Oncology Group): 0-2
2. Histologic documentation of invasive duct or lobular adenocarcinoma of the breast
3. If neoadjuvant chemotherapy was NOT administered: pathologic T1-3, N1-2 following definitive surgery
4. If neoadjuvant chemotherapy was administered, pathology from the definitive surgery must confirm pathologic T1-3, N1-2 disease and also meet one of the following criteria:

   Clinical T1-3, N1-2 or Pathologic confirmation of axillary nodal involvement at presentation (ie, before neoadjuvant therapy) based on any of the following: Positive fine-needle aspiration (FNA), Positive core needle biopsy.
5. Complete resection of known breast disease by one of the following surgeries Lumpectomy with axillary lymph node dissection with no more than 12 resected lymph nodes.

Mastectomy and axillary lymph node dissection with no more than 12 resected lymph nodes.

5- ER(estrogen-receptor), PR (progesterone-receptor), and HER2(human epidermal growth factor receptor 2) testing performed on the primary breast tumor; when applicable, testing must have been performed before receiving neoadjuvant chemotherapy.

6-Margins of the resected specimen must be histologically free of invasive tumor and ductal carcinoma in situ (DCIS) as determined by the pathologist.

7-The surgical wound should be completely healed without any signs of infection.

8-Interval between the last surgery for breast cancer or the completion of adjuvant chemotherapy and study enrollment must be ≤ 56 days (ie, a maximum of 8 weeks).

9-If adjuvant chemotherapy is received there should be at least 10 days gap between the last day of chemotherapy and the enrollment in the study to avoid skin toxicity.

10-Women of child-bearing potential must agree to use a medically accepted form of pregnancy prevention for the duration of study treatment 11-Ability to understand and willingness to sign the consent form written in Arabic

Exclusion Criteria:

1. Patients with surgical margins less than or equal to 2mm.
2. Patients with axillary dissection of more than 12 lymph nodes due to high incidence of arm lymphedema.
3. Women with Huge pendulous breast.
4. Patients with bad breast conservative surgery ( Surgery that impair the cosmetic outcome before starting radiotherapy).
5. T4 tumors including inflammatory breast cancer.
6. Known definitive clinical or radiologic evidence of metastatic disease.
7. Patients re operated for microscopic positive margins after definitive surgery.
8. Previous radiation therapy for the currently diagnosed breast cancer prior to study enrollment
9. History of ipsilateral or contralateral breast or thoracic radiotherapy for any condition
10. History of ipsilateral or contralateral axillary surgery for any condition
11. History of lymphedema involving the ipsilateral or contralateral arm at present or at any time in the past
12. Active collagen vascular disease, specifically dermatomyositis with a creatine phosphokinase (CPK) level above normal or with an active skin rash, systemic lupus erythematosis, or scleroderma.
13. Pregnancy or breastfeeding
14. Second primary cancer.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-02 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Locoregional recurrence | 5 years
  Tumor locoregional recurrence is defined as: Any newly suspicious skin change/s or palpable lymph node in the irradiated area (compared to baseline photo and clinical examination of this area) that is/are pathologically proved to be locoregional tumor recurrence.
  Suspicious skin change/s and palpable lymph node from baseline photo and baseline clinical examination of the irradiated area will be monitored at 3 months throughout 5 years following the completion of radiotherapy in the two study arms to detect the incidence and time of locoregional recurrence.
Cosmetic outcomes | 5 years
  Aesthetic evaluation of the irradiated breast will be through 3 methods. Patient questionnaire (Subjective evaluation), Harvard score for breast cosmoses (Observer evaluation) and a computer soft ware that calculate the configuration difference between treated and non treated breast. Upon evaluation, each of the three methods will acquire a point ranging from 0 to 3 (poor to excellent cosmetic outcome respectively). The points of the three methods will be added yielding a score ranging from 0 to 9. Score 0-2, 3-4, 5-6 and 7-9 mean poor, fair, good and excellent cosmoses respectively.
  The cumulative incidence of changes in breast cosmoses from baseline for every patient will be assessed every year (as described above) through out the 5 years (Time frame of the study) following the completion of radiotherapy in the two study arms. By the end of the five years the aesthetic evaluation for each patient will be through calculating the average of her 5 years score.
Arm lymph edema. | 5 years
  To evaluate the cumulative incidence of lymph edema during the 5 years following completion of hypofractionated radiation treatment [ Time Frame: 5 years ] Incidence of lymphedema defined as ≥ 10% increase in arm circumference over baseline circumference compared to the contralateral arm measured every 6 months from the time of initiation of hypofractionated irradiation of breast and regional nodes through 5 years following the completion of radiation therapy in 2 study groups.
Health economic perspectives | 5 years
  The economic perspectives for the public health: (Time frame 5 years). Cost effective analysis of each treatment plan will be evaluated at the end of 5 years through calculation of the cost-effectiveness ratio = Cost of intervention / Health effect produced.
  The cost of intervention = the sum of (Cost of medical staff time, drugs and equipment maintenance during the 5 years time frame). (The cost of intervention during the 5 years time frame will be used for calculations).
  The health effect produced will be years of local control (Number of years the patient lived without any pathological evidence of local recurrence). (The mean years of local control during the 5 years time frame will be used for calculations).
  The treatment program with the less cost effectiveness ratio will be recommended for treating patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Ellithy, Phd, Principal Investigator — Ain Shams University
Locations (1):
- Mahmoud Ellithy, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No